CLINICAL TRIAL: NCT06690658
Title: Self-Practicing Upper Body Exercises with a Robotic Trainer System in the Physical Therapy Department: a Feasibility Study
Brief Title: Self-Practicing Upper Body Exercises with a Robotic Trainer System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, shirley handelzalts, Principal investigator, Loewenstein Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0007-23-LOE
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-11

CONDITIONS: Robot Assisted Therapy; Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thirty people with lower limb orthopedic injury or lower limb amputation (Other): Participants will be asked to fill pre-experiments questionnaires. Each patient will be assigned a unique number before the first session, which they will use to log into the system.
  The patient together with the physical therapist will schedule the time for the patient to self-practice with the system, 3 times per week for 3 weeks, 30 min each session. A training session begins with the robot introducing itself, and the participant sits in front of the robot. The robot will demonstrate upper body exercises and will provide verbal instructions and feedback. The participant will be asked to follow the robot's demonstration and simultaneously perform the exercise. When completing the training program, the users will be asked to fill in questionnaires. After each session, the participant will be asked to rate his perceived rate of exertion using the Borg scale (0 to 10 scale) on the robot's screen and will be offered to start the training session from the beginning.
  Interventions: Device: incorporating robotic system for upper body physical training of people with lower limb orthopedic condition

INTERVENTIONS:
Device: incorporating robotic system for upper body physical training of people with lower limb orthopedic condition — A training session begins with the robot introducing itself, and the participant sits in front of the robot. The robot will demonstrate upper body exercises and will provide verbal instructions and feedback (e.g, number of successful repetitions, motivational). At the beginning of the session, the participant will be asked to follow the robot's demonstration and simultaneously perform the exercise. At the end of each exercise, the robot will provide feedback. If the participant successfully performed ten repetitions of the required exercise in the demonstration time allocated, positive feedback will be provided. Resistance (strengthening) exercises for the upper body include lifting weights, working with resistance bands in different directions involving the upper extremity and trunk. Flexibility exercises include upper extremity and trunk stretching.

SUMMARY:
Studies suggest that older adults undergoing inpatient rehabilitation have relatively low levels of physical activity. Moreover, people with lower limb orthopedic conditions undergoing inpatient rehabilitation may be particularly vulnerable to the consequences of low physical activity because of the mobility limitations.

The study focuses on examining the feasibility of incorporating robotic system for upper body physical training of people with lower limb orthopedic condition undergoing inpatient rehabilitation. Using robotic coaches can be a complementary method to promote the participation and motivation of people with lower limb orthopedic conditions undergoing inpatient rehabilitation.

Aims:

The overall aim of the study is to assess the user experience and feasibility of incorporating robotic system for upper body physical training of people with lower limb orthopedic injury/condition undergoing inpatient rehabilitation. Our specific aims are:

1. To assess the acceptability and suitability of the training (i.e., training attendance and engagement; adherence to training protocol; time on task; satisfaction and enjoyment of the training)
2. To document unexpected adverse events during training.
3. To assess the resources and ability to manage and implement the training (i.e., administrative capacity, technology and equipment needs and training).

DETAILED DESCRIPTION:
The training will be conducted in a designated area in the physical therapy hall. After completing the consent form, participants will be asked to fill pre-experiments questionnaires including demographic information as well as details about their profession, education, and other personal attributes, Negative Attitude towards Robots (NARS) questionnaire, and Technology Adoption Propensity (TAP) Questionnaire. The physical therapist, together with the patient, will choose specific strengthening and flexibility exercises from multiple options according to participant's ability and training goals. The physical therapist will explain about the system and how it works prior to the beginning of the session. In addition, to ensure that each patient can access their customized training, each patient will be assigned a unique number before the first session, which they will use to log into the system The patient together with the physical therapist will schedule the time for the patient to self-practice with the system, 3 times per week for 3 weeks. A training session begins with the robot introducing itself, and the participant sits in front of the robot. The robot will demonstrate upper body exercises and will provide verbal instructions and feedback (e.g, number of successful repetitions, motivational). At the beginning of the session, the participant will be asked to follow the robot's demonstration and simultaneously perform the exercise. At the end of each exercise, the robot will provide feedback. If the participant successfully performed ten repetitions of the required exercise in the demonstration time allocated, positive feedback will be provided. Resistance (strengthening) exercises for the upper body include lifting weights, working with resistance bands in different directions involving the upper extremity and trunk. Flexibility exercises include upper extremity and trunk stretching. Rest breaks will be provided as needed during the session. Participants will be able to stop the training at any time. During the training, the system will collect data regarding the success of the exercises in excel files without any identifiable data. When completing the training program, the users will be asked to fill in questionnaires. During all training sessions, a physical therapist will be present in the room to provide guidance and supervision, ensuring that the exercises are performed correctly and do not induce pain or fatigue. The therapist will also review the kinematic data collected in each session to monitor progression and adjust the program (such as increasing or decreasing exercise difficulty). After each session, the participant will be asked to rate his perceived rate of exertion using the Borg scale (0 to 10 scale) on the robot's screen and will be offered to start the training session from the beginning.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ Age
* stable clinical and metabolic state
* ability to sit without back support independently
* ability to understand research instructions.

Exclusion Criteria:

* A contraindication to perform active upper extremity movements
* Severe pain that limits the ability to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Training attendance | From enrollment to end of treatment at 3-4 weeks

SECONDARY OUTCOMES:
Time on task (in minutes) | From enrollment to end of treatment at 3-4 weeks.
The physical activity enjoyment scale | From enrollment to end of treatment at 3-4 weeks.
User Experience Questionnaire - Short Version (UEQ-S) | From enrollment to end of treatment at 3-4 weeks.
Almere Model scale | From enrollment to end of treatment at 3-4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Hospital, Raanana, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes